CLINICAL TRIAL: NCT02483442
Title: D-dimer Testing,Tailored to Clinical Pretest Probability to Reduce the Use of CT Pulmonary Angiography in Suspected Pulmonary Embolism: A Management Study (The Pulmonary Embolism Graduated D-dimer [PEGeD] Study)
Brief Title: D-dimer Testing Tailored to Clinical Pretest Probability in Suspected Pulmonary Embolism
Acronym: PEGeD
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: OCOG-2014-PEGeD
Record Dates: First submitted 2015-06-18; First posted 2015-06-29 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No CT Pulmonary Angiography: Low Clinical Pretest Probability with D-dimer < 1000 ug/L and Moderate Clinical Pretest Probability with D-dimer < 500ug/L
- CT Pulmonary Angiography Required: Low Clinical Pretest Probability with D-dimer > or = 1000ug/L and Moderate Clinical Pretest Probability with D-dimer > or = 500 ug/L and High Clinical Pretest Probability

SUMMARY:
Prospective, multicentre, cohort study assessing a diagnostic management strategy for suspected Pulmonary Embolism with independent central adjudication of outcomes

DETAILED DESCRIPTION:
This is a prospective, multi-centre, cohort study that will assess a new diagnostic management strategy for suspected Pulmonary Embolism (inpatients and outpatients). The new diagnostic strategy is designed to reduce the use of imaging tests for Pulmonary Embolism, particularly Computed Tomography Pulmonary Angiogram, by excluding Pulmonary Embolism with combinations of Clinical Pretest Probability and D-dimer results in a higher proportion of patients. The safety of this management strategy will be established by demonstrating a very low rate of proximal Deep Vein Thrombosis or Pulmonary Embolism during 90 days of follow-up in patients who had anticoagulant therapy withheld in response to negative diagnostic testing. Diagnostic test utilization will be assessed. All clinical outcomes will be adjudicated by a central independent adjudication committee that will be blind to initial D-dimer measurements and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Patients (either outpatients or inpatients) with clinically suspected Pulmonary Embolism.

Exclusion Criteria:

1. Age less than 18 years.
2. Treated with full-dose anticoagulation for ≥ 24 hours before D-dimer was measured.
3. Major surgery (general or spinal anesthesia) in the past 21 days.
4. Result of the D-dimer assay that will be used to manage the patient in the study is known before Clinical Pretest Probability was done.
5. Computed Tomography Pulmonary Angiogram or Ventilation Perfusion Scan was performed:

   1. before Clinical Pretest Probability was documented, or
   2. in a patient with Low Clinical Pretest Probability and a D-dimer level <1,000 ug/L (or equivalent), or
   3. in a patient with Moderate Clinical Pretest Probability and a D-dimer level <500 ug/L (or equivalent).
6. Computed Tomography of the chest with contrast will be performed for another reason (e.g. to assess for malignant disease or aortic dissection), and would be performed even if Pulmonary Embolism is excluded by Clinical Pretest Probability and D-dimer testing.
7. Ongoing need for anticoagulant therapy.
8. Life expectancy less than 3 months.
9. Geographic inaccessibility which precludes follow-up.
10. Known pregnancy.
11. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients (either outpatients or inpatients) with clinically suspected Pulmonary Embolism.
Sampling Method: Non-Probability Sample
Enrollment: 2038 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with confirmed symptomatic proximal Deep Vein Thrombosis or Pulmonary Embolism | 90 Days (+ or - 7days)
  Proximal Deep Vein Thrombosis includes thrombosis confined to the calf vein trifurcation but not isolated more distal Deep Vein Thrombosis. Pulmonary Embolism does not include isolated sub-segmental abnormalities on Computed Tomography Pulmonary Angiography.

SECONDARY OUTCOMES:
Number of patients with bleeding | 90 days (+ or - 7days)
  Major and minor bleeding
Number of patient Deaths | 90 days (+ or - 7days)
  All deaths and cause specific deaths
Number of patients with Venous Thromboembolism | 90 days (+ or - 7days)
  Venous Thromboembolism, including events that do not satisfy the primary outcome (e.g. isolated distal Deep Vein Thrombosis or subsegmental Pulmonary Embolism) but that are confirmed by the adjudication committee.

CONTACTS AND LOCATIONS:
Overall Officials: Clive Kearon, MD, Principal Investigator — McMaster University
Locations (9):
- Canada (9):
  - University of Alberta Hospital, Edmonton, Alberta
  - HHS- Hamilton General Hospital, Hamilton, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - HHS - McMaster University Medical Centre, Hamilton, Ontario
  - Juravinski Hospital, Hamilton, Ontario
  - London Health Sciences, London, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sherbrooke University Hospital, Sherbrooke, Quebec
  - Jewish General Hospital, Montreal

REFERENCES:
- [Derived] Kearon C, de Wit K, Parpia S, Schulman S, Afilalo M, Hirsch A, Spencer FA, Sharma S, D'Aragon F, Deshaies JF, Le Gal G, Lazo-Langner A, Wu C, Rudd-Scott L, Bates SM, Julian JA; PEGeD Study Investigators. Diagnosis of Pulmonary Embolism with d-Dimer Adjusted to Clinical Probability. N Engl J Med. 2019 Nov 28;381(22):2125-2134. doi: 10.1056/NEJMoa1909159. PMID 31774957